CLINICAL TRIAL: NCT02266719
Title: Clinical Outcomes and Radiation Safety After Endovascular Repair of Complex Aortic Aneurysms Using Fenestrated and Branched Devices
Brief Title: Clinical Outcomes and Radiation Safety After Endovascular Repair of Complex AAAs Using Fenestrated- Branched Devices
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Carlos H Timaran, Associate Professor of Surgery, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G140108
Record Dates: First submitted 2014-10-06; First posted 2014-10-17 (Estimated); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Aortic Aneurysm, Abdominal; Thoracic Aneurysm
Keywords: Aortic Aneurysm, Abdominal [C14.907.055.239.075]; Thoracic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aortic Aneurysm, Thoracic; Aortic Aneurysm

STUDY DESIGN:
Intervention Model Description: The study is divided in three groups, as follows:
  Patients with complex abdominal aortic aneurysms including, juxtarenal, suprarenal and type IV thoracoabdominal aneurysms will be enrolled in the fenestrated-CMD group.
  Patients with type I-III throacoabdominal aneurysms will be enrolled in the type I-III TAAAs groups and will be eligible for custom-made/ off-the-shelf branched devices.
  Patients with high surgical risk with aortic arch aneurysms treated by patient-specific stent-grafts with one to three inner branches or a scallop.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Fenestrated CMD cohort (Experimental): Patients enrolled in this arm will be implanted with the custom made fenestrated device. The device is aimed to treat complex abdominal aortic aneurysms including juxtarenal, suprarenal and type IV thoracoabdominal aneurysms.
  Interventions: Device: Fenestrated CMD
- Type I - III TAAA cohort (Experimental): Patients enrolled in this arm will be implanted with the custom made/ off-the-shelfp branched devices. The device is aimed to treat type I-III TAAAs.
  Interventions: Device: Type I - III TAAA
- Arch cohort (Experimental): Patients enrolled in this arm will be implanted with patient-specific stent-grafts with one to three inner branches or a scallop.
  Interventions: Device: Arch cohort

INTERVENTIONS:
Device: Fenestrated CMD — The CMD that will be used in this IDE is structurally the same as the commercially available Zenith Fenestrated AAA Endovascular Graft.
  In general, the Zenith® Fenestrated AAA Endovascular Graft is a modular system constructed of full- thickness woven polyster fabric sewn to self-expanding stainless steel z-stents with braided polyster and monofilament polypropylene sutures. In this study, fenestrated grafts with usually up to 4 fenestrations may be used.
  Device implantation will be performed using standardized endosvacular techniques used in the treatment of abdominal aortic aneurysms.
  Other Names: Cook Zenith® Fenestrated CMD
  Arms: Fenestrated CMD cohort
Device: Type I - III TAAA — Device implantation will be performed using standardized endosvacular techniques used in the treatment of abdominal aortic aneurysms. Devices will be implanted in patients with type I-III thoracic abdominal aneurysms.
  The branches in this study will be constructed as internal/external cuffs, axially oriented and caudally or cranially directed, as necessary . Branch position will be determined by the anatomic location of the target vessels using a consistent craniocaudal and circumferential cuff position.
  Other Names: CMD-off-the-shelf branched devices-
  Arms: Type I - III TAAA cohort
Device: Arch cohort — Arch branched devices may be designed using one of two configurations: (1) Zone 0 device with two inner antegrade branches for the innominate artery and the left common carotid artery with or without a retrograde left subclavian artery branch and (2) Zone 1-2 device with a single retrograde subclavian artery branch with double or triple wide scallop for the left common carotid artery. These devices are designed for a of proximal landing/fixation zone of at least 20 mm of healthy aortic segment or a previous graft.
  Other Names: Zenith Arch Branch Device
  Arms: Arch cohort

SUMMARY:
The purpose of this study is to assess the clinical outcomes and radiation of the use of off-the-shelf and custom-made devices (CMDs) for the endovascular repair of juxtarenal, suprarenal, thoracoabdominal and arch aortic aneurysms in patients having appropriate anatomy. The study consists of three cohorts. The first 2 cohorts are the continuation of the current IDE study. The first cohort is aimed to assess the use of custom-made devices (CMDs) for the endovascular repair of juxtarenal, suprarenal and type IV thoracoabdominal aortic aneurysms in standard and high-risk patients having appropriate anatomy (Fenestrated-CMD cohort). The second cohort (Type I-III thoracoabdominal cohort) includes standard and high-risk patients with type I- III thoracoabdominal aneurysms that require the use of branched/fenestrated CMDs, or, in selected cases, the Zenith Thoracoabdominal Branch (Zenith® t-Branch™) device. Finally, the third cohort (the Arch cohort) will include 25 high-risk patients with aortic arch aneurysms treated by patient-specific stent-grafts with one to three inner branches or a scallop

DETAILED DESCRIPTION:
This study is a prospective, single center, non-randomized, triple-cohort study. For the Fenestrated-CMD cohort a total of 350 patients will be enrolled. For the type I-III thoracoabdominal cohort, a total of 250 patients will be enrolled. For the Arch cohort, 25 patients will be enrolled. CMDs will be used primarily. Off-the-shelf devices will be used in urgent cases and when the waiting period for design and manufacturing of a CMD may not be considered acceptable. Staged endovascular repair will be used for type I, II and III TAAAs and for concurrent arch and TAAAs, unless the condition of the patient requires a single stage endovascular repair. A separate subgroup analysis of patients undergoing procedures with off-the-shelf devices will be performed.

ELIGIBILITY:
General Inclusion Criteria

A patient is deemed suitable for inclusion in the study if the patient has at least one the following:

1. Juxtarenal or suprarenal AAA, type I-IV thoracoabdominal aortic aneurysms or aortic arch aneurysms or dissections with diameter ≥5.0 cm in diameter or 2 times the normal aortic diameter;
2. Aneurysm with history of growth ≥0.5 cm/year;
3. Saccular aneurysm with aortic diameter greater than 1.5 times the normal aortic diameter that is deemed to be at risk for rupture based upon physician interpretation.
4. Patients that are not eligible for treatment with commercially available endografts.
5. Presence of concomitant thoracoabdominal and aortic arch aneurysm meeting one of the above-mentioned criteria.

General Exclusion Criteria

A patient must be excluded from the clinical investigation if any of the following are true:

1. Age <18 years;
2. Life expectancy <2 years;
3. Pregnant, breast-feeding, or planning on becoming pregnant within 60 months;
4. Inability or refusal to give informed consent by the patient or a legally authorized representative;
5. Unwilling or unable to comply with the follow-up schedule;
6. Prior surgical or interventional procedure within 30 days of the anticipated date of the fenestrated procedure, with the exception of planned staged procedures to provide access for repair (e.g. staged iliac conduit, thoracic endovascular aortic aneurysm repair for proximal aneurysms, elephant trunk repair), to facilitate the procedure by allowing open reparation of a target artery not amenable to revascularization with the investigational device, such us an internal iliac artery, subclavian artery or visceral artery with early bifurcation, tortuosity or occlusive disease preventing successful placement and alignment side stents, or to treat proximal aortic aneurysms.
7. Participation in another clinical or device trial, with the exception of observational studies, participation in another investigational endovascular endograft protocol, percutaneous aortic valve protocol, or concomitant clinical trials designed to evaluate medical therapy strategies to reduce perioperative risk during fenestrated-branched endovascular repair, including risks of renal dysfunction, contrast-induced nephropathy, neurologic, spinal cord or cardiac complications, and/or use of advanced imaging to reduce radiation exposure during implantation of these devices. Participation in investigational device trials not encompassed by the IDE protocol should be performed remotely from the fenestrated/branched repair (>30 days). Participation in medical therapy trial or advanced imaging trial designed to improve peri-operative outcomes or to reduce radiation exposure of fenestrated/branched endografts may be concurrent with the IDE study. Examples include therapy directed to reduce rates of spinal cord injury, stroke and contrast-induced nephropathy associated with implantation of fenestrated-branched stent-grafts or advanced imaging trials designed to reduce radiation exposure during repair.
8. Patients with ruptured aortic aneurysm requiring urgent or emergent repair, with the exception of patients with contained, stable ruptures with anatomy suitable for an off-the-shelf design.
9. Patients who meet anatomical criteria for commercially available aortic stent-grafts according to proposed instructions for use of these devices.

Medical Exclusion Criteria

Patients must be excluded from the study if any of the following conditions are true:

1. Known sensitivities or allergies to stainless steel, nitinol, polyester, solder (tin, silver), polypropylene, urethane or gold
2. History of anaphylactic reaction to contrast material that cannot be adequately pre-medicated
3. Leaking or ruptured aneurysm associated with hypotension
4. Uncorrectable coagulopathy
5. Mycotic aneurysm or patients with evidence of active systemic infection.
6. History of connective tissue disorder (e.g. vascular Ehlers Danlos, Marfan syndrome), with the exception of those patients who had prior open surgical aortic replacement or endovascular repair, where a surgical graft or an endograft would serve as landing zone for the investigational endograft, those who are deemed prohibitive risk for open repair or connective tissue disorders with no vascular effects (e.g. non-vascular types of Ehlers Danlos).
7. Body habitus that would inhibit x-ray visualization of the aorta and its branches.

Anatomical Exclusion Criteria

Patient must be excluded from the study if any of the following is true:

1. Inadequate femoral or iliac access compatible with the requirements of the required delivery system.
2. Inability to perform a temporary or permanent open surgical or endovascular iliac conduit for patients with inadequate femoral/iliac access.
3. Absence of a landing aortic segment in the distal thoracic aorta above the diaphragmatic hiatus with:

   1. A diameter measured outer to the outer wall greater than 42 mm or less than 19 mm;
   2. Parallel aortic wall with >20% diameter change and with significant calcification and/or thrombus in the selected area of the seal zone.
4. Visceral anatomy not compatible with the investigational device due to excessive occlusive disease or small size not amenable to stent graft placement.
5. Unsuitable distal iliac arterial fixation site and anatomy:

   1. Common iliac artery fixation site diameter measured outer wall to outer wall on a section image (CT)< 8.0 mm with inability to perform surgical conduit.
   2. Iliac artery diameter measured outer wall to outer wall on a sectional image (CT) > 21 mm at distal fixation site, with inability to perform open internal iliac artery revascularization or iliac branch stent graft or custom iliac extension with fenestration.
   3. Iliac artery distal fixation site <10 mm in length.
   4. Inability to preserve at least one hypogastric artery.

For patients in the type I-III TAAA cohort, the intended use criteria are the same for both the fenestrated/branched CMD vs the off-the-shelf device. The CMD will preferably be used, unless an urgent repair is indicated or the waiting period for design or manufacturing of the CMD is considered unacceptable.

Additional anatomical inclusion criteria for aortic arch devices

1. Proximal aortic fixation zone:

   1. Native aorta or surgical graft
   2. Diameter: 20-42mm
   3. Proximal neck length ≥ 20mm
   4. Ascending aortic length ≥50mm
   5. Must occur distal to coronary arteries and any coronary artery bypass grafts that are considered patent and necessary for proper cardiac perfusion
2. Distal aortic fixation zone:

   1. Native aorta or surgical graft
   2. Diameter: 20-42mm
   3. Distal neck length ≥20mm
   4. Distal fixation will be obtained with stent-grafts in a staged repair
3. Supra-aortic trunk (brachiocephalic) vessels

   1. The arch branch device will typically have two or three branches with additional modifications to the design that allows for a single branch or combination of branch and scallop if a customized version is required. An extra-anatomic bypass graft may be done in conjunction (or in a staged fashion) with the procedure, as required. For the two-branch design, the vessels most commonly incorporated will be the innominate artery and left common carotid artery. However, the innominate artery may be coupled with the left subclavian artery in the setting of a bovine arch whereby the flow to the left carotid would come from a left subclavian to carotid bypass. Similarly, the left carotid and subclavian artery may be branched, or simply one vessel branched should specific anatomic limitations exist. In such a situation, multiple extra-anatomic bypasses may be necessary. A design with a single subclavian retrograde branch and scallop to the left carotid artery may be used to extent the landing zone to Zone 1. Finally, a design with two antegrade inner branches for the innominate and left common carotid, and one retrograde inner branch for the left subclavian artery may be used in select cases. Thus, the inclusion criteria are defined for each artery, yet any combination of arteries may be used for a repair.

   i. Innominate artery

1. Native vessel or surgical graft

2. Diameter: 8-22mm

3. Length of sealing zone ≥10mm

4. Acceptable tortuosity

ii. Left (or right) common carotid artery

1. Native vessel or surgical graft
2. Diameter 6-16mm
3. Length of sealing zone ≥10mm
4. Acceptable tortuosity

iii. Left (or right) subclavian artery

1. Native vessel or surgical graft
2. Diameter: 5-20mm
3. Length of sealing zone ≥10mm
4. Acceptable tortuosity

4. In the setting of an aortic dissection the following criteria must exist:

1. Access into the true lumen from the groin and at least one supra-aortic trunk vessel
2. A sealing zone in the target aorta (or surgical graft) that is proximal to the primary dissection, such that a stent-graft would be anticipated to seal off the dissection lumen
3. A sealing zone in the target supra-aortic trunk vessels that is distal to the dissection, anticipated to seal off the dissection lumen, or surgically created
4. A true lumen size large enough to deploy the device and still gain access into the target branches

   5. In the setting of more distal disease, the repair may be coupled with a thoracoabdominal branched device, infrarenal device, and/or internal iliac branch device.

   6. Iliac anatomy must allow for the delivery of the arch branch device which is loaded within a 20F-24F sheath. Conduits to the iliac vessels or aorta may be used if deemed necessary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 625 (Estimated)
Dates: Start 2014-12-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate safety endovascular treatment of juxtarenal, suprarenal, thoracoabdominal and arch aortic aneurysms using fenestrated/branched investigational devices. | 30 days
  Primary safety will be defined as the proportion of subjects who experience a major adverse event (MAE) at 30-days or during hospitalization if this exceeds 30 days.
Evaluate effectiveness endovascular treatment of juxtarenal, suprarenal, thoracoabdominal and arch aortic aneurysms using fenestrated/branched investigational devices. | 12-months
  For primary effectiveness endpoint, treatment success will be analyzed as the proportion of patients to achieve treatment success at 12-months.

SECONDARY OUTCOMES:
Rate of Grafts deployed at intended site with successful and patent stenting of target vessels (technical success) | 30 days
  Technical success is defined as successful access of the aneurysm site and deployment of endovascular graft in the intended location. The endovascular graft and all vessels targeted with fenestrations must be patent at the time of deployment completion as evidenced by intraoperative angiography.
Number of Major adverse events | 5 years
  Major adverse events are defined as the occurrence of any of the following: death, aneurysm rupture, or conversion to open surgical repair; Q wave myocardial infarction (MI); cardiac ischemia requiring intervention; renal failure requiring dialysis; bowel obstruction or bowel ischemia requiring intensification of medical therapy or surgical therapy; aorto-enteric fistula; stroke; paralysis.
Number of participants with adverse events from the use of bare metal stents as a measure of safety | 5 years
  When bare metal balloon expandable or self-expandable stents are required to be used distally to covered stents, target vessel events (kink, stenosis or occlusion) will be analyzed separately at 30 days, 6 months and annually up to five years.

OTHER OUTCOMES:
Rate of complications not considered as major (Secondary safety endpoints) | 30 days
  Other Major adverse events such as paraplegia and paraparesis, stroke and specific mortality.
Rate of successful procedures and treatment in terms of device integrity (Secondary effectiveness endpoints) | 5 years
  Treatment success and procedure success. Endograft integrity will be evaluated within this outcome measurement.
Number of participants with adverse events from radiation exposure as a measure of tolerability. | 5 years
  Skin changes secondary to radiation exposure will be evaluated within this outcome measurement.
Rate of major adverse events in patients treated with low profile devices (Safety for low profile devices) | 5 years
  Safety will be defined as the proportion of subjects who experience a major adverse event for patients treated with low profile devices.
Rate of procedures with successful access of aneurysm site and deployment of low profile devices with patent stenting of target vessels (Effectiveness for low profile devices) | 5 years
  Effectiveness is defined as technical success (successful access of the aneurysm site and deployment of endovascular graft in the intended location. The endovascular graft and all vessels targeted with fenestrations must be patent at the time of deployment completion as evidenced by intraoperative angiography)of low profile devices use.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Mesnard T, Huang Y, Schanzer A, Timaran CH, Schneider DB, Mendes BC, Eagleton MJ, Farber MA, Parodi FE, Gasper WJ, Beck AW, Sweet MP, Zetterval SL, Lee A, Oderich GS; United States Aortic Research Consortium. Multicenter Prospective Evaluation of Patient Radiation Exposure During Fenestrated-Branched Endovascular Aortic Repair: A Ten-year Experience. Ann Surg. 2025 Feb 18. doi: 10.1097/SLA.0000000000006676. Online ahead of print. PMID 39963789
- [Derived] Oderich GS, Huang Y, Harmsen WS, Tenorio ER, Schanzer A, Timaran CH, Schneider DB, Mendes BC, Eagleton MJ, Farber MA, Gasper WJ, Beck AW, Sweet MP, Lee WA; United States Aortic Research Consortium. Early and Late Aortic-Related Mortality and Rupture After Fenestrated-Branched Endovascular Aortic Repair of Thoracoabdominal Aortic Aneurysms: A Prospective Multicenter Cohort Study. Circulation. 2024 Oct 22;150(17):1343-1353. doi: 10.1161/CIRCULATIONAHA.123.068234. Epub 2024 Jul 11. PMID 38989575
- [Derived] Finnesgard EJ, Beck AW, Eagleton MJ, Farber MA, Gasper WJ, Lee WA, Oderich GS, Schneider DB, Sweet MP, Timaran CH, Simons JP, Schanzer A; United States Aortic Research Consortium. Severity of acute kidney injury is associated with decreased survival after fenestrated and branched endovascular aortic aneurysm repair. J Vasc Surg. 2023 Oct;78(4):892-901. doi: 10.1016/j.jvs.2023.05.034. Epub 2023 Jun 16. PMID 37330702
- [Derived] Aucoin VJ, Motyl CM, Novak Z, Eagleton MJ, Farber MA, Gasper W, Oderich GS, Mendes B, Schanzer A, Tenorio E, Timaran CH, Schneider DB, Sweet MP, Zettervall SL, Beck AW; U.S. Aortic Research Consortium. Predictors and outcomes of spinal cord injury following complex branched/fenestrated endovascular aortic repair in the US Aortic Research Consortium. J Vasc Surg. 2023 Jun;77(6):1578-1587. doi: 10.1016/j.jvs.2023.01.205. Epub 2023 Apr 13. PMID 37059239
- [Derived] Timaran LI, Timaran CH, Scott CK, Soto-Gonzalez M, Timaran-Montenegro DE, Guild JB, Kirkwood ML. Dual fluoroscopy with live-image digital zooming significantly reduces patient and operating staff radiation during fenestrated-branched endovascular aortic aneurysm repair. J Vasc Surg. 2021 Feb;73(2):601-607. doi: 10.1016/j.jvs.2020.05.031. Epub 2020 May 27. PMID 32473339
- [Derived] Timaran DE, Knowles M, Ali T, Timaran CH. Fenestrated endovascular aneurysm repair among octogenarians at high and standard risk for open repair. J Vasc Surg. 2017 Aug;66(2):354-359. doi: 10.1016/j.jvs.2016.11.064. Epub 2017 Feb 16. PMID 28216359
- [Derived] Timaran DE, Soto M, Knowles M, Modrall JG, Rectenwald JE, Timaran CH. Safety and effectiveness of total percutaneous access for fenestrated endovascular aortic aneurysm repair. J Vasc Surg. 2016 Oct;64(4):896-901. doi: 10.1016/j.jvs.2016.03.444. Epub 2016 May 27. PMID 27237404